CLINICAL TRIAL: NCT03160937
Title: Neurodynamic Mobilization and Foam Rolling in Delayed-onset Muscle Soreness in a Healthy Adult Population: a Randomized Controlled Clinical Trial
Brief Title: Neurodynamic Mobilization and Foam Rolling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Daniel Muñoz-Garcia, PhD, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSEULS-PI-009/2013
Record Dates: First submitted 2017-05-13; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Exercise-induced Muscle Damage; Movement Disorders; Nerve Pain
Keywords: pain
MeSH Terms: conditions — Movement Disorders; Neuralgia; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: a single NM treatment session on Delayed Onset Muscle pain (DOMS) and to compare them with those of one foam roller (FR) session
Who Masked: Outcomes Assessor
Masking Description: One single evaluator who was blinded to the group assignments performed all tests that occurred 5 minutes prior to and 5 minutes after the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy Foam (Experimental): The subjects included rolled the foam roller down their quadriceps using short kneading-like motions until it was just above their patellae, and then rolled it back to its initial position in one fluid motion. The subjects repeated this motion for 1 min, rested for 30 s, and then repeated it again for 5 sets
  Interventions: Other: Manual therapy
- Manual therapy Nerve (Active Comparator): The subjects was positioned lying on his/her side with a pillow underside leg (without fully flexing it) and the cervical and thoracic spines flexed. The investigator flex the knee and the hip extended and then put it back to its initial position in one fluid motion. The subjects repeated this motion for 1 min, rested for 30 s, and then repeated it again for 5 sets
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — The subjects repeated this motion for 1 min, rested for 30 s, and then repeated it again for 5 sets.

SUMMARY:
The purpose of this study was to assess the acute effects of a single NM treatment session on DOMS and to compare them with those of one foam roller (FR) session. Following the damaging plyometric exercise bout, the participants were randomly assigned in a counter-balanced fashion to either a FR or NM treatment group; treatments were administered 48-h post-exercise. The dependent variables were recorded before the exercise, 48-h post-exercise before treatment, and immediately post-treatment.

DETAILED DESCRIPTION:
Currently, the foam-rolling massage is often used by athletes from many sports. However, there are a few studies on the effects of foam-rolling massage and they have conflicting results regarding the improvements in ROM and muscular performance. In contrast, neurodynamic mobilization (NM) is a manual therapy method used to assess and treat neuromuscular disorders. It includes gliding techniques and tensile techniques. Gliding techniques or "sliders" are intended to produce a sliding movement between neural structures and adjacent nonneural tissues. NM has been shown to reduce pain and soreness and improve ROM. However, no studies have investigated its effects after exercise-induced muscle soreness or DOMS.

ELIGIBILITY:
Inclusion Criteria:

* All subjects were moderately active (Category 2) as assessed by the International Physical Activity Questionnaire (IPAQ) questionnaire (Craig et al., 2003).
* None of the subjects had a recent history of intensive training, heavy eccentric resistance, or plyometric exercise, and all subjects were free from musculoskeletal disorders in the last year.
* All subjects were asked to refrain from unaccustomed exercise during the experimental period, and the subjects abstained from all medications and dietary supplements during the experimental period and between testing sessions.

Exclusion Criteria:

* Sedentary
* patients with pain

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Pain | 1 minute after treatment
  the numeric pain-rating scale (NPRS)

SECONDARY OUTCOMES:
Leg dynamometer measurements | 2 minutes after treatment
  Leg strength
Surface electromyography (sEMG) | 5 minutes after treatment
  EMG of quadriceps muscle

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Muñoz, PhD, Principal Investigator — Centro Universitario La Salle

IPD SHARING:
Plan to Share IPD: No